CLINICAL TRIAL: NCT04276662
Title: An Open-label, Single-dose Study to Assess the Pharmacokinetics of DS-3201b In Subjects With Hepatic Impairment
Brief Title: Study of Single-dose DS-3201b in Participants With Hepatic Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS3201-A-U106
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Hepatic Impairment
Keywords: Hepatic Impairment; DS-3201b; Enhancer of zeste homolog (EZH) inhibitor

STUDY DESIGN:
Intervention Model Description: Phase 1, open-label, parallel design, single-dose PK study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1: Mild hepatic impairment (Experimental): Participants who have mild hepatic impairment as assessed by National Cancer Institute Organ Dysfunction Working Group (NCI-ODWG) criteria.
  Interventions: Drug: DS-3201b
- Cohort 2: Moderate hepatic impairment (Experimental): Participants who have moderate hepatic impairment as assessed by National Cancer Institute Organ Dysfunction Working Group (NCI-ODWG) criteria.
  Interventions: Drug: DS-3201b
- Cohort 3: Healthy participants (Experimental): Healthy participants who have normal hepatic function with sex, age (±10 years [y]), and weight (±20%) matching with the mild and moderate hepatic impairment cohorts.
  Interventions: Drug: DS-3201b

INTERVENTIONS:
Drug: DS-3201b — 1 dose of 50 mg DS-3201b

SUMMARY:
This is a Phase 1, open-label, parallel design, single-dose pharmacokinetic (PK) study to assess the safety, tolerability, and PK of a single dose of 50 mg of DS-3201b in participants with normal and impaired hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants 18 years to 75 years of age (inclusive), with a body mass index (BMI) of 18 kg/m^2 to 40 kg/m^2 (inclusive) and body weight between 50 kg and 120 kg (inclusive) at Screening.
* Female participants who are of non-childbearing potential must be:
* Surgically sterile (ie, bilateral tubal ligation or removal of both ovaries and/or uterus at least 6 months prior to dosing, or Essure® with hysterosalpingogram [documentation to confirm tubal occlusion 12 weeks [wk] after procedure]).
* Naturally postmenopausal (spontaneous cessation of menses) for at least 24 consecutive months prior to dosing, confirmed by follicle stimulating hormone (FSH) or estradiol testing.
* Female participants of childbearing potential with proper means of hormonal and nonhormonal or barrier contraceptive methods; all female participants must have negative pregnancy tests at Screening and Check-in. Female participants must be using proper contraceptive means for at least 1 month prior to Screening. Acceptable means of contraceptive methods include sexual abstinence, vasectomy of male partner, intrauterine device, barrier methods like female condom, diaphragm or cervical cap, spermicide, hormonal contraceptives, or any combination of above. Female participants who normally abstain from sexual activity may be recruited provided that they agree to use a condom and spermicide should they become sexually active at any time during the study and for 90 days post dose. Male partners should also be informed to use a condom during this study period. Participants with hepatic impairment should consult with their primary care physician about using any oral contraceptive options (eg, would a combination of hormonal contraception and barrier contraceptive methods be allowed by the physician).
* Male participants must agree to use a condom and spermicide during sexual intercourse until 90 days post dose or must have had a vasectomy and must be willing not to donate sperm until 90 days post dose. Female partners of male participants should be informed of additional barrier contraceptive during this time and may use barrier and/or hormonal contraceptive methods under the conditions described below. Participants with hepatic impairment should consult with their primary care physician about hormonal contraceptive options for their partner. Participants should use both hormonal and barrier methods of contraception for themselves and their partner.
* Participants must agree to refrain from donation of blood from 56 days prior to Screening, plasma from 2 wk prior to Screening, and platelets from 6 wk prior to Screening. Participants must also agree to refrain from donation of blood until 56 days after the end of study.
* All participants must be willing to refrain from consuming grapefruit/grapefruit juice, Seville oranges, and pomegranates/pomegranate juice 10 days before the study drug is given on Day 1 until End-of-Study.
* Participants with hepatic impairment are required to have:

  1. Documented history of chronic liver disease diagnosed by ultrasonography, computed tomography scan, liver biopsy, or magnetic resonance imaging or history of chronic (>6 months) hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
  2. Hepatic impairment as assessed by NCI-ODWG classification 2

     Mild hepatic impairment as assessed by:
     * Total bilirubin (Tbil) ≤upper limit of normal (ULN) and AST >ULN, or
     * Tbil >1 to 1.5 × ULN (not due to Gilbert's syndrome)

     OR

     Moderate hepatic impairment as assessed by:
     * Tbil >1.5 to 3 × ULN (not due to Gilbert's syndrome)
  3. Physical examination findings that are normal or not clinically significant and clinical laboratory evaluations with normal limits or not clinically significant deviations, with exception of findings that in the opinion of the investigator are consistent with the participant's hepatic impairment
  4. Clinical stability in the opinion of the investigator. No evidence of active HBV and/or new or acute HCV infection within the preceding 6 months.
* Estimated creatinine clearance (CrCl) ≥60 mL/min by Cockcroft-Gault equation at Screening and Check-in

Exclusion Criteria:

* Clinically relevant abnormal history, physical findings, electrocardiogram, or laboratory values at the Screening assessment that could interfere with the objectives of the study or the safety of the participant
* Participants with primary biliary cirrhosis or primary sclerosing cholangitis
* Participants with history of Gilbert's syndrome
* Use of any drugs or substances known to be moderate/strong inhibitors or inducers of CYP3A4 and 3A5 enzymes or P-glycoprotein (P-gp) inhibitors within 14 days or 5 half-lives, if known, of the drugs or substances, whichever is greater, prior to study drug administration
* Receipt of any prescribed or over-the-counter (OTC) systemic, herbal (including St John's wort), or topical medication within 14 days of study drug administration, or any expectation of requiring use of such medication while participating in the study is prohibited
* Presence or history of clinically severe adverse reaction to any drug
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (with the exception of appendectomy, hernia repair, and/or cholecystectomy)
* History of any cancer, except non-melanoma skin cancer, or resected non-metastatic cancer with no evidence of disease accepted by the Investigator and Sponsor medical monitor
* A positive drugs of abuse screen from a urine ethanol test (unless the drug is medically prescribed by a licensed health care provider) or alcohol breath test at Screening or at Check-in on Day -2 or a participant who will not agree to smoke ≤10 cigarettes or equivalent per day from Screening up to Enrollment, and is unable to be restricted to ≤5 cigarettes per day and for 6 hours post dose during their period of residence in the clinical unit
* Concomitant use of medications known to affect the elimination of serum creatinine (eg, trimethoprim or cimetidine) and inhibitors of renal tubular secretion (eg, probenecid) within 14 days or 5 half-lives, if known, of the drugs, whichever is greater, prior to study drug administration
* History or presence of an abnormal electrocardiogram, which, in the investigator's opinion, is clinically significant and/or a QT interval corrected for heart rate using Fridericia's formula ≥450 milliseconds (ms) and ≥470 ms for healthy male and female participants, respectively, and >500 ms for subjects with hepatic impairment at Screening
* Consumption of alcohol- and caffeine-containing beverages within 72 hours prior to Check-in and during confinement
* History of moderate to heavy alcohol use defined as consumption of more than 28 units of alcohol per week for males or 14 units of alcohol per week for females, where 1 unit of alcohol equals one-half pint of beer, 4 ounces (oz) of wine, or 1 oz of spirits, or significant history of alcoholism or drug/chemical abuse within the last 2 years
* Positive serology for hepatitis B surface antigen (HBsAg) and HCV (healthy participants), hepatitis A virus (HAV) immunoglobulin M, or anti-human immunodeficiency virus (HIV) Type 1 and Type 2 (participants)
* Loss of more than 450 mL blood during the 3 months before the trial (eg, as a blood donor)
* Current enrollment in or have not yet completed at least 30 days or 5 elimination half-lives, whichever is longer, since receiving an investigational device or product, or receipt of other investigational agents within 30 days of DS-3201b
* In the opinion of the investigator, history of a clinically significant illness within 4 wk prior to administration of study drug
* Women of childbearing potential without proper nonhormonal or barrier contraceptive measures and women who are pregnant or breastfeeding. Male and female participants may be excluded from the study if the primary investigator at the site forbids specific methods of contraception they are using.
* Start of any new medication or any changes to a current dosage within 14 days prior to study drug administration excluding approved oral contraceptives

Additional Exclusion Criteria for Matched Healthy Participants:

* Any clinically relevant abnormality identified on the physical examination, electrocardiogram, vital signs, or laboratory tests at Screening
* Liver function (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase (ALP) of liver origin, gamma glutamyltransferase [GGT], and Total bilirubin [TBil]) test results above the ULN at Screening and during Enrollment on Day -2 are exclusionary. If transaminase levels are >2 × ULN at Screening the participant will be excluded and cannot be rescreened

Additional Exclusion Criteria for Participants with Hepatic Impairment:

* Participants with active stage 3 or stage 4 encephalopathy
* Fluctuating or rapidly deteriorating hepatic function as indicated by recent history or worsening of clinical and/or laboratory signs of hepatic impairment as judged by the investigator
* Participants with known portal hypertension and/or had shunting procedures done

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
Analysis of Pharmacokinetic Parameter: Maximum Concentration of DS-3201a (Cmax) | 1 to 10 days postdose
  Cmax is the maximum concentration of DS-3201a in plasma
Analysis of Pharmacokinetic Parameter: Area under the concentration-time curve from time zero to time of last measurable concentration of DS-3201a (AUClast) | 1 to 10 days postdose
  AUClast is the area under the concentration-time curve from time zero to time of last measurable concentration of DS-3201a in plasma
Analysis of Pharmacokinetic Parameter: Area under the concentration-time curve up to infinity of DS-3201a (AUCinf) | 1 to 10 days postdose
  AUCinf is the area under the concentration-time curve up to infinity of DS-3201a in plasma
Analysis of Pharmacokinetic Parameter: Time to reach maximum concentration of DS-3201a (Tmax) | 1 to 10 days postdose
  Tmax is the time to reach maximum concentration of DS-3201a in plasma
Analysis of Pharmacokinetic Parameter: Apparent total body clearance of DS-3201a (CL/F) | 1 to 10 days postdose
  CL/F is the apparent total body clearance of DS-3201a in plasma
Analysis of Pharmacokinetic Parameter: Apparent volume of distribution of DS-3201a (Vz/F) | 1 to 10 days postdose
  Vz/F is the apparent volume of distribution of DS-3201a in plasma
Analysis of Pharmacokinetic Parameter: Terminal elimination half-life of DS-3201a (t1/2) | 1 to 10 days postdose
  t1/2 is the terminal elimination half-life of DS-3201a in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (3):
- United States (3):
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - Worldwide Clinical Trials, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/